CLINICAL TRIAL: NCT05614271
Title: A Prospective Cohort Study Exploring the Associations Between Chronic Postsurgical Pain and Postoperative Cognitive Dysfunction After Elective Knee or Hip Arthroplasty
Brief Title: Chronic Postsurgical Pain, Postoperative Cognitive Dysfunction and Resilience
Acronym: ArthroCaP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: The McMaster Institute for Research on Aging (MIRA) (Unknown); Michael G. DeGroote Institute for Pain Research and Care (IPRC) (Unknown)
Responsible Party: Principal Investigator, Maura Marcucci, Assistant Professor, Department of Health Research Methods, Evidence and Impact and Department of Medicine, McMaster University
Other Study IDs: 13598
Record Dates: First submitted 2022-10-28; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Postoperative Cognitive Dysfunction; Chronic Post Operative Pain; Satisfaction, Patient; Coping Behavior
Keywords: Older adults; Total knee arthroplasty; Total hip arthroplasty; Postoperative cognitive dysfunction; chronic postsurgical pain
MeSH Terms: conditions — Postoperative Cognitive Complications; Pain, Postoperative; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
"Brain damage" and "memory loss" are main concerns of people undergoing surgery. In fact, many older people undergoing different types of non-cardiac surgeries (including orthopedic surgeries) present a significant decline in their cognition (i.e. the way people use their brain to think, take action, make decision, and remember) 1 year after surgery. This is called postoperative cognitive dysfunction (POCD), and is significantly more frequent (as many as 30% of patients aged 65 or older) than what we would expect in non-surgical patients with similar age and comorbidities. Causes and mechanisms of POCD are poorly understood. Pain after surgery is also very frequent and can persist for a long time (i.e. persistent postsurgical pain, PPSP), requiring chronic medications including narcotics. Knee surgery is more often offered as a treatment in older patients with osteoarthritis, who often come to surgery after a long history of pain and impaired mobility, and who often experience PPSP. The investigators proposed to conduct a study in 200 people 55 years old or older (expected age range 55-85) who are undergoing their elective knee surgery, to evaluate the association between PPSP (and its treatment) and POCD. How cognition can interfere with resilience (coping strategies and expectations), which are also thought to influence the persistence of pain, satisfaction, and functional recovery after surgery, will also be explored. Patients will be enrolled before their surgery and followed over time, to collect data on their social and clinical characteristics, measure copying/expectations before and after surgery, and assess pain and pain medications, satisfaction and functional recovery, and cognitive performance. The study will also explore hypotheses of possible mechanisms underlying the association between PPSP and POCD, and will include interviews with a subset of the participants to explore lived experiences of pain, mobility and aging, including resilience, expectations and satisfaction with surgery.

DETAILED DESCRIPTION:
The specific study objectives are to: 1- explore the association of CPSP, pain management (opioid use), and patient satisfaction, with postoperative cognitive dysfunction (POCD), measured both as change in the Montreal Cognitive Assessment (MoCA), and through a neuropsychological test battery, 2- explore whether postoperative cognitive changes are associated with changes in neurogenesis correlates and in neurotrophic factors levels, and whether this association is mediated by changes in pain, mobility, and satisfaction, and 3- explore the association between coping strategies/expectations as measured by the Somatic Preoccupation and Coping (SPOC) questionnaire and cognitive function, and in particular the relationship between changes in SPOC and cognitive changes from preoperative to 4-6 weeks after surgery.

Investigators will recruit 150 patients, 50 years or older scheduled for knee or hip arthroplasty 1-2 weeks before surgery (baseline) and collect information about their socio-demographics data, comorbidities, frailty, anxiety, pain, and pain medications. The SPOC questionnaire is administered at baseline and repeated at 4-6 weeks after surgery. CPSP (presence and severity) and satisfaction with surgery are measured at 3, 6, and 12 months. Cognitive / neuropsychological assessments will be administered at baseline, and 4-6 weeks, 6 months, and 12 months after surgery. Blood samples for serum and RNA expression analysis of biomarkers will be longitudinally collected with the same timeline.

ELIGIBILITY:
Inclusion Criteria:

1. aged 50 years or older,
2. scheduled for elective TKA or THA for osteoarthritis
3. able to provide informed consent.

Exclusion Criteria:

1. known history of dementia,
2. unavailability of tablet or computer with an internet connection for remote assessment,
3. patient unable to interact with a tablet or computer due to language, visual, or hearing impairment, or any severely limited mobility of the upper limb joints, OR
4. patient unable to understand spoken or written English.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 50 years or older undergoing elective total knee arthroplasty (TKA) or total hip arthroplasty (THA) for osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative cognitive dysfunction (binary outcome) | 6 and 12 months postoperative
  defined as a >=2 point decline in MoCA scores.

SECONDARY OUTCOMES:
Changes in the Mnemonic Similarity Test scores | 4-6 weeks and 6 and 12 months
  Participants are first engaged in an encoding phase then a subsequent recognition test with a 3-choice response; exact repetitions of earlier items, lures (similar but not identical to earlier items), and novel foils. During the test, participants are asked to identify each item as "Old," "Similar," or "New". The lure discrimination index (which measures mnemonic discrimination) is calculated as the difference between the rate of "Similar" responses given to the lure items minus "Similar" responses given to the foils. Typically, 'normal' aging is associated with a decline in mnemonic discrimination (identifying lure objects that are similar to memory set objects as "similar") with preserved recognition memory (identifying repeated memory set objects as "old"). The MST version used in the study is a validated modified online version of MST adapted to increase the efficiency of the test.
Changes in the Visual Paired Associates Learning (PAL) test | 4-6 weeks and 6 and 12 months
  A computer task that assesses visual memory and new learning by testing a participant's memory for object location pairs. Boxes are displayed on the screen and are opened in a randomized order. One or more of them will contain a pattern. The patterns are then displayed in the middle of the screen, one at a time, and the participant must touch the box where the pattern was originally located. If the participant makes an error, the patterns are represented by their locations. The difficulty increases throughout the test. The average accuracy across the last two completed levels will be analyzed
Changes in the Rapid serial Visual Presentation (RVP) test | 4-6 weeks and 6 and 12 months
  A white box is shown in the centre of the screen, inside which digits from 2 to 9 appear in a pseudo-random order, at the rate of 100 digits per minute. Participants are requested to detect target sequences of digits (for example, 2-4-6, 3-5-7, 4-6-8). When the participant sees the target sequence they must respond by selecting the button in the centre of the screen as quickly as possible. The level of difficulty varies with either one- or three-target sequences that the participant must watch for at the same time. The average accuracy throughout the task will be analyzed.
Changes in the Stroop color word color interference task CWIT | 4-6 weeks and 6 and 12 months
  CWIT has the standard color naming, word reading, and color-word interference trials,in addition to additional trial requiring the examinee to switch between inhibitory and non-inhibitory responses. Process measures enable assessment of general difficulties. Condition 1: Color Naming, Condition 2: Word Reading, Condition 3: Inhibition, Condition 4: Inhibition/ Switching requires adequate naming speed, reading speed, verbal inhibition, and cognitive flexibility.and Scores will include the time needed to complete each condition, the number of errors and the number of self-corrected errors
Changes in the N-back test | 4-6 weeks and 6 and 12 months
  Participants are shown a series of numbers on the screen and are asked to enter the number they saw two numbers ago. The outcome measures are correct detection and reaction times.

CONTACTS AND LOCATIONS:
Overall Officials: Maura Marcucci, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT05614271/Prot_SAP_000.pdf